CLINICAL TRIAL: NCT07099391
Title: ALTITUDE - ALTernating Induction Therapies to Achieve Undetectable Disease Endpoints: A Phase 1/2 Alternating Dara-RVd/Teclistamab-RVd in Transplant Eligible Standard-risk Newly Diagnosed Multiple Myeloma
Brief Title: A Study of Dara-RVd and Teclistamab-RVd in People With Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-288
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; ALTITUDE; Dara-RVd; Teclistamab-RVd; Memorial Sloan Kettering Cancer Center; 24-288
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I (Experimental): The phase 1 part of the study evaluates the safety and toxicity of Tec-RVd
  Interventions: Drug: Dara-RVd; Drug: Tec-RVd
- Phase II, Stage 1 (Experimental): The phase II part of the study evaluates MRD negativity (MRD-) rate of alternating Dara-RVd/Tec-RVd after 6 cycles of induction therapy. If 4 or less participants achieve a MRD- after 6 cycles evaluation the trial will be stopped. If 5 or more participants accomplish a MRD- the trial will move on to stage 2
  Interventions: Drug: Dara-RVd; Drug: Tec-RVd
- Phase II, Stage 2 (Experimental): The phase II part of the study evaluates MRD negativity (MRD-) rate of alternating Dara-RVd/Tec-RVd after 6 cycles of induction therapy.
  Interventions: Drug: Dara-RVd; Drug: Tec-RVd

INTERVENTIONS:
Drug: Dara-RVd — This study is a phase 1/2 study design of alternating 6 cycles of Dara-RVd/Tec-RVd induction therapy
Drug: Tec-RVd — This study is a phase 1/2 study design of alternating 6 cycles of Dara-RVd/Tec-RVd induction therapy

SUMMARY:
The purpose of this study is to find out whether Tec-RVd (teclistamab, lenalidomide, bortezomib, and dexamethasone) after 3 treatment Cycles of Dara-RVd (daratumumab, lenalidomide, bortezomib, and dexamethasone) is a safe treatment for people with newly diagnosed multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

1. Documented multiple myeloma satisfying the International Myeloma Working Group (IMWG) diagnostic criteria36 (evidence of myeloma defining event attributed to underlying plasma cell disorder) with measurable disease defined as:

   1. Clonal plasma cells in the bone marrow ≥ 10% or presence of a biopsy proven plasmacytoma
   2. Measurable disease within the past 4 weeks defined by any of the following:

      * IgG myeloma: Serum monoclonal protein ≥ 1.0 g/dL or urine monoclonal protein ≥ 200 mg/24 hr; or
      * IgA, IgM, IgD, IgE multiple myeloma: serum M-protein ≥ 0.5 g/dL or urine monoclonal protein ≥ 200 mg/24 hr; or
      * Light chain multiple myeloma: Involved serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum free kappa/lambda light chain ratio
      * Measurable plasmacytomas seen on imaging (≥ 1 lesion that has a single diameter ≥ 2 cm). If this is the primary marker of measurable disease, patients will need a biopsy at screening.
      * Bone marrow plasma cells ≥ 30% as determined by CD138 immunohistochemistry staining.
2. Standard risk multiple myeloma - excluding patients with high risk cytogenetic abnormality (HRCA) according to the IMS/IMWG 2024 Consensus Definition:

   1. TP53 mutation and/or del(17p) with cancer clonal function (CCF) >20% by analyses conducted on CD138+ purified cells
   2. t(4;14), t(14;16), or t(14;20) co-occurring with +1q (gain/amp 1q) and/or del(1p)
   3. Monoallelic del(1p32) with +1q or biallelic del(1p32)
   4. High Beta-2 microglobulin (>5.5 mg/dL) with normal creatinine (<1.2 mg/dL)
3. Newly diagnosed patient considered a candidate for high-dose chemotherapy and autologous stem cell transplant

   a. For patients who received one complete cycle of Dara-RVd at MSK, patients can enter treatment at cycle 2 at the discretion of treating investigator and PI
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Have adequate organ and hematologic function:

   1. Hemoglobin ≥ 7.5 g/dL (prior RBC transfusion or recombinant human erythropoietin use is permitted);
   2. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L (G-CSF use is permitted);
   3. Platelet count ≥ 75 x 109/L
   4. Creatinine Clearance ≥ 30 ml/min. CrCl can be measured or estimated using Cockcroft-Gault method, MDRD, or CKD-EPI formula
   5. Total bilirubin ≤ 2 x ULN (≤ 3 x ULN if documented Gilbert's syndrome);
   6. AST ≤ 2.5 x ULN;
   7. ALT ≤ 2.5 x ULN
7. All study participants must be able to tolerate one of the following thromboprophylaxis strategies: aspirin, low molecular weight heparin or warfarin (coumadin) or alternative anti-coagulant.
8. All study participants must be able to tolerate one of the following thromboprophylaxis strategies: aspirin, low molecular weight heparin or warfarin (Coumadin), or direct-acting oral anticoagulants (DOACs).
9. All study participants must be registered into the mandatory REMS® program and be willing and able to comply with the requirements of REMS®, including compliance with contraception methods (Appendix A).

Exclusion Criteria:

1. Patients who have received > 1 cycle of prior treatment or concurrent systemic therapy for multiple myeloma (excluding corticosteroids or radiation therapy). For patients who received one complete cycle of Dara-RVd at MSK, patients can enter treatment at cycle 2 at the discretion of treating investigator and PI
2. Patients with diagnosis of plasma cell leukemia, primary light chain amyloidosis, monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), Waldentröm's macroglobulinemia
3. History of another active primary malignancy within 2 years prior to enrollment, except for adequately treated basal cell carcinoma or squamous cell skin cancer or carcinoma in situ.
4. Significant, uncontrolled comorbid conditions that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in the study. Examples include, but are not limited to

   1. Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal.
   2. Moderate or severe persistent asthma within the past 2 years or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
   3. Infiltrative pulmonary disease
   4. Active autoimmune disease requiring systemic immunosuppressive therapy within 6 months before start of study treatment. Exception of vitiligo, type 1 diabetes, and prior autoimmune thyroiditis that is currently euthyroid
   5. Disabling psychiatric conditions (e.g., alcohol or drug abuse)., severe dementia, or altered mental status
   6. Known history of human immunodeficiency virus (HIV)
   7. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]).

   i. Subjects with resolved infection (i.e., subjects who are HBsAg negative with antibodies to total hepatitis B core antigen [anti-HBc] with or without the presence of hepatitis B surface antibody [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded.

   ii. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of HBV vaccination, do not need to be testing for HBV DNA by PCR.

   h. Seropositive for hepatitis C i. Except in the setting of a sustained virologic response [SVR], defined as a viremia at least 12 weeks after completion of antiviral therapy.

   i. Clinically significant cardiac disease, including: i. Myocardial infarction within 6 months before enrollment, or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV) ii. Uncontrolled cardiac arrhythmia
5. Pregnant or lactating patients
6. Unwilling to give written, informed consent, unwilling to participate, or unable to comply with the protocol for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2029-07-24 (Estimated); Study Completion 2029-07-24 (Estimated)

PRIMARY OUTCOMES:
Phase I: Toxicity | up to 4 months
  Evaluate the safety and toxicity of Tec-RVd for Phase I participants by the number of Dose Limiting Toxicities experienced within the DLT window
Phase II: MRD Negativity | up to 6 months
  The primary endpoint is MRD negativity (MRD-) rate upon completion of 6 cycles of alternating Dara-RVd with Tec-RVd.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Korde, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org